CLINICAL TRIAL: NCT04971928
Title: A Phase 1, Open-label, Single-Dose Study to Evaluate the Pharmacokinetics of GSK3228836 in Adults With Hepatic Impairment and Healthy Matched Control Participants (B-Assured)
Brief Title: Phase 1 Study of GSK3228836 Pharmacokinetics in Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205871
Record Dates: First submitted 2021-06-22; First posted 2021-07-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Hepatitis B
Keywords: GSK3228836; Hepatitis B; Child-Pugh B (CP-B) cirrhosis; Child-Pugh A (CP-A) cirrhosis; Pharmacokinetics; B-Assured
MeSH Terms: conditions — Hepatitis B; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants with Moderate (CP-B) hepatic impairment (Experimental)
  Interventions: Drug: GSK3228836
- Participants with Mild (CP-A) hepatic impairment (Experimental)
  Interventions: Drug: GSK3228836
- Healthy participants (Experimental)
  Interventions: Drug: GSK3228836

INTERVENTIONS:
Drug: GSK3228836 — GSK3228836 will be administered

SUMMARY:
This is a Phase 1, open-label, parallel-group study to evaluate the pharmacokinetics of GSK3228836 in participants with Child-Pugh B (CP-B) cirrhosis (moderate hepatic impairment), Child-Pugh A (CP-A) cirrhosis (mild hepatic impairment) and participants with normal hepatic function as healthy control.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >50 Kilogram (kg) and body mass index (BMI) within the range 19 to 40 Kilogram per square meters (kg/m2) (inclusive)
* Capable of giving signed informed consent.
* Child-Pugh B cirrhosis (moderate hepatic impairment; Part 1) or Child-Pugh A cirrhosis (mild hepatic impairment; Part 2) or a healthy control participant based on a medical evaluation including medical history, physical examination (PE), laboratory tests.

Exclusion Criteria:

* Diagnosed or suspected hepatocellular carcinoma.
* History of malignancy within the past 5 years except for cancers that are cured by surgical resection (e.g., skin cancer).
* History of vasculitis or presence of symptoms and signs of potential vasculitis or history/presence of other diseases that may be associated with vasculitis condition.
* Unstable cardiac function or high blood pressure that is not controlled (based on the investigator's discretion).
* Any other medical condition which, in the judgment of the investigator and Medical Monitor, could jeopardize the integrity of the data derived from that participant or the safety of the participant.
* Participants who have taken or are currently taking any therapies not allowed by the protocol.
* A positive test for human immunodeficiency virus (HIV) antibody.
* History of sensitivity to GSK3228836 or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from time zero (pre-dose) extrapolated to infinite time [AUC(0-infinity)] | Up to Day 50 post-dose
Maximum observed concentration (Cmax) | Up to Day 50 post-dose

SECONDARY OUTCOMES:
AUC from time zero (pre-dose) to 24 hours [AUC(0-24)] | Up to 24 hours post-dose
AUC from time zero (pre-dose) to 168 hours [AUC(0-168)] | Up to 168 hours post-dose
Plasma concentration of GSK3228836 on Day 8 | Day 8 post-dose
Apparent terminal phase half-life (t1/2) | Up to Day 50 post-dose
Apparent clearance (CL/F) | Up to Day 50 post-dose
Time of occurrence of Cmax (Tmax) | Up to Day 50 post-dose
Apparent terminal phase volume of distribution (Vz/F) | Up to Day 50 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com